CLINICAL TRIAL: NCT01024088
Title: Prospective Study on Swallowing/Breathing Interactions in Severe Guillain Barre Syndrome.
Acronym: DGVSB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P061016 -CRC 06040
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2011-02

CONDITIONS: Tetraplegia; Respiratory Failure
Keywords: Guillain Barré syndrome; Swallowing disorders; Respiratory failure
MeSH Terms: conditions — Quadriplegia; Respiratory Insufficiency; Guillain-Barre Syndrome; Deglutition Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GBS PATIENT
- CONTROL

SUMMARY:
To estimate, in a longitudinal and not invasive way, in patients with SGB at respiratory risk, the function of respiratory muscles and that of the upper airways muscles by investigating the force of the tongue, the gulp, and the breath during the sleep to be able to detect bulbar impairment and establish correlations enter the various parameters to estimate better the interactions between the dysfunction of the respiratory muscles and that upper airways muscles and so determine the risk acute respiratory failure.

DETAILED DESCRIPTION:
Context: the syndrome of Guillain Barré ( SGB) is the first causes of extensive paralysis of medical origin in industrial nations. A third of these patients going to require mechanical invasive ventilation during their stay in ICU. This population of ventilated presents the strongest risk of infectious respiratory patient complications and death. The respiratory impairment is a progressive weakness of inspiratory and expiratory muscles. The monitoring of the respiratory muscular infringement is usually made by the repeated measure of vital capacity and the maximal respiratory pressures. The occurrence of bulbar impairment is an aggravating element entailing dysfunction of the upper airways muscles detected often late in front of aspiration. Besides the arisen of sleep apneas was never sought in this context. This dysfunction of the upper airways muscles could be more detected prematurely by objectivizes measures of them performances.

Method: longitudinal observational and in a one center study. The respiratory impairment will be estimated by the measure of the vital capacity, maximal respiratory pressures and of the debit of cough. The existence of a bulbar infringement will be sought by the measure of the force of the tongue, an objective measure of gulp performances and a polysomnographic recording.

Criterion of selection: patient admitted in ICU with GBS and respiratory risk. Number of patients, centre: 40 patients admitted in the intensive care unit of the hospital RAYMOND POINCARE and 20 controls.

Duration of the study: 24 months Perspectives: better anticipate acute respiratory failure and the indication of an invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Guillain Barré Syndrome
* Presenting a risk of mechanical ventilation(breakdown): presence of 2 among the following 5 criteria

  * Deficit evolving for less than 7 days
  * Impossibility to stand up
  * Impossibility to raise the head
  * ineffective Cough
  * Vital capacity< 60 %

Exclusion Criteria:

* MAJOR confusions of gulp (spontaneous) at admittance
* Respiratory distress syndrome and intubation at admission buccal dental lesions
* Not membership to a regime of Social Security (beneficiary or legal successor)
* Patient under guardianship or custody

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient admitted in ICU with GBS and respiratory risk
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Correlation between respiratory failure and bulbar dysfunction during ICU stay | 24 MONTHS

SECONDARY OUTCOMES:
Number of aspiration pneumonia | 24 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: David Orlikowski, PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- hôpital Raymond Poincaré, Garches, France